CLINICAL TRIAL: NCT07192991
Title: Neuroendocrine Carcinomas: Patient Journey And Treatment Outcomes In Latin America
Acronym: NECTARINE
Status: Not yet recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Boehringer Ingelheim (Industry); Grupo Argentino de Investigación Clínica en Oncología (Unknown); Grupo de Estudios Clínicos Oncológicos Peruano (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 1324
Record Dates: First submitted 2025-02-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Carcinomas; Lung Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor block: Formalin-Fixed Paraffin-Embedded collected from 2014 onwards.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with extra-pulmonary neuroendocrine carcinoma: Patients with Extrapulmonary Neuroendocrine Carcinoma (EP-NEC), diagnosed between August 2014 and August 2024.
  Interventions: Other: Observational study
- Patients with pulmonary neuroendocrine carcinoma: Patients with Large-cell neuroendocrine carcinoma (LCNEC) or mixed and patients with Small Cell Lung Cancer (SCLC) or mixed, diagnosed between August 2014 and August 2024.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
This observational, retrospective study aims to understand the treatment patterns and outcomes of patients with pulmonary and extra-pulmonary neuroendocrine carcinomas (NEC) in Latin America (Brazil, Mexico, Argentina, and Peru). The research will collect data from medical records to analyze factors like patient demographics, diagnosis methods, tumor characteristics, treatment approaches, and disease progression. The study is non-interventional, meaning patient care will follow standard clinical practice, with data gathered via an electronic system.

DETAILED DESCRIPTION:
Currently, there is a hypothesis that there is not enough evidence to fully understand the patient journey and accurately determine the clinical outcomes of neuroendocrine carcinomas (NEC) in Latin America. A better understanding of this landscape, including its unique regional aspects, could lead to improved patient care.

To address this gap, this observational, retrospective, non-interventional study aims to describe treatment patterns and outcomes for patients with both pulmonary and extra-pulmonary NEC in Latin America. Eligible patients diagnosed with either form of NEC will be included, and data will be collected from medical records at selected sites across Brazil, Mexico, Argentina, and Peru.

Data to be retrieved include but are not limited to age at diagnosis, gender, ECOG at diagnosis, stage (TNM), resources used for primary diagnosis (imaging, upfront surgery etc.), primary site, tumor size and grade, setting of initial treatment (reference center vs community hospital), type of initial surgical approach, data of anti-cancer treatments (including (neo)adjuvant and advanced settings) and relapse and/or progression/death. Data regarding anti-cancer treatments (including (neo)adjuvant and advanced settings), as well as radiotherapy use will also be recorded.

As this project is non-interventional, patients will still receive treatment and clinical assessments for extra-pulmonary and pulmonary NEC as determined by their attending physician, according to the standard of care and routine clinical practice at each site. No visits are demanded by the study, but for those required for the consent process whenever determined by the local ethics committee. Patient source data will be taken from the patient's medical records and reported by means of an electronic data capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosed between August 2014 and August 2024 with one of the following:
* Extrapulmonary Neuroendocrine Carcinoma (EP-NEC)
* Large-cell neuroendocrine carcinoma (LCNEC) or mixed
* Small Cell Lung Cancer (SCLC) or mixed
* Adequate and accessible medical records for data collection
* Tumor block collected from 2014 onwards

Exclusion Criteria:

* Patients with active, concurrent malignancies at the time of NEC diagnosis, except for non-invasive cancers like basal cell carcinoma or squamous cell carcinoma of the skin, or in situ cervical cancer.
* Patients or their legal representatives unwilling or unable to provide informed consent (if needed per ethics committee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extra-pulmonary neuroendocrine carcinoma (EP-NEC) and patients with pulmonary neuroendocrine carcinoma (SCLC or LCNEC) from Brazil, Mexico, Argentina and Peru.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patterns of Initial Cancer Treatment: number of participants treated within vs. outside high-volume sites and associated treatment characteristics | Throughout the study period, an average of 24 months
  Treatment patterns will be analyzed descriptively using tables and graphs to illustrate the distribution of patients receiving initial cancer treatment within versus outside high-volume treatment centers. Key characteristics of the initial treatment will be assessed.
Event-free survival (EFS) | Throughout the study period, an average of 24 months
  defined as time from diagnosis until relapse, death, or definitive failure of treatment strategy that implicates failure of curative-intent treatment [for patients treated with curative intent]. Participants who are lost to follow up or reach the study end will be censored at their last date of contact.
Time to treatment failure (TTF) | Throughout the study period, an average of 24 months
  in first and second-line: defined as time from first dose of treatments until date of discontinuation of treatment for any reason, including progression of disease, treatment toxicity, and death. Participants who are lost to follow up or reach the study end will be censored at their last date of contact
Progression-free survival (PFS) | Throughout the study period, an average of 24 months
  defined as time from treatment initiation until progression or death [for patients treated with palliative intent]. Participants who are lost to follow up or reach the study end will be censored at their last date of contact.
Overall survival | Throughout the study period, an average of 24 months
  [according to disease stage/setting], defined as time from initial diagnosis until date of death from any cause. Participants who are lost to follow up or reach the study end will be censored at their last date of contact.
Frequency of DLL-3 immunohistochemistry expression | After the end of recruitment, an average of 1 year
  Rate of patients with DLL3 expression in extra-pulmonary and pulmonary NEC by IHC [stratified by tumor primary site]

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Simões Pimenta Riechelmann, Principal Investigator — Latin American Cooperative Oncology Group; Vladmir Cláudio Cordeiro de Lima, Principal Investigator — Latin American Cooperative Oncology Group